CLINICAL TRIAL: NCT00544687
Title: A Phase I, Single-Center, Randomized, Vehicle and Active-Controlled Study to Assess and Compare the Atrophy-Causing Potential of Topical CRx-191 Formulations in Healthy Volunteers
Brief Title: Phase I Study of Topical CRx-191 in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zalicus (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRx-191-002; EudraCT Number: 2006-005903-33
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Skin; Atrophy; CRX-191; mometasone furoate; nortriptyline hydrochloride; Skin Thickness in Normal Healthy Volunteers
MeSH Terms: conditions — Atrophy | interventions — Mometasone Furoate; Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): CRx-191 (0.1% mometasone furoate + 0.05% nortriptyline HCl)
  Interventions: Drug: CRx-191
- 2 (Experimental): CRx-191 (0.1% mometasone furoate + 0.1% nortriptyline HCl)
  Interventions: Drug: CRx-191
- 3 (Active Comparator): 0.1% mometasone furoate
  Interventions: Drug: mometasone furoate
- 4 (Active Comparator): 0.1% nortriptyline HCl
  Interventions: Drug: nortriptyline HCl
- 5 (Active Comparator): Karison® Creme (clobetasol-17-propinate 0.05%)
  Interventions: Drug: Karison® Creme
- 6 (Placebo Comparator): Vehicle (placebo)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CRx-191 — topical (mometasone furoate + nortriptyline HCl)
  Arms: 1; 2
Drug: mometasone furoate — topical mometasone furoate
  Arms: 3
Drug: nortriptyline HCl — topical nortriptyline HCl
  Arms: 4
Drug: Karison® Creme — topical Karison® Creme (clobetasol-17-propinate 0.05%)
  Arms: 5
Drug: Vehicle — topical (placebo)
  Arms: 6

SUMMARY:
CRx-191 is a proprietary synergistic combination drug candidate being evaluated by CombinatoRx for topical psoriasis therapy. CRx-191 was identified via a proprietary screening assay for novel drug combinations demonstrating enhanced inhibition of tumor necrosis factor- alpha and interferon-gamma release, cytokines that are implicated in the pathogenesis of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily give written informed consent
* Subject must be at least 18 years of age
* Subject must have healthy skin on which reddening can be easily recognized in the area of the test fields
* The physical examination must be without disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the study
* Sexually active females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective medically accepted contraceptive regimen; systemic contraceptive (combined oral contraceptive, implant, injection), or safe intrauterine device (IUD)
* Written informed consent obtained

Exclusion Criteria:

* Acne, suntan, eczema, hyper- or hypopigmentation, or tattoos in the test fields
* Dark skinned persons whose skin color prevents ready assessment of skin reactions
* Cardiac disease including recent myocardial infarction, any degree of heart block or other cardiac arrhythmias and valvular heart disease
* Mania
* Narrow angle glaucoma
* Hyperthyroidism by medical history, TSH < LLN, or receiving thyroid medication
* Severe liver disease (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) laboratory values that exceed 1.5x ULN)
* Inflammatory dermatoses (e.g. atopic dermatitis, psoriasis), bacterial, viral, or fungal skin infections; facial rosacea
* Active varicella, tuberculosis, syphilis or post-vaccine reactions
* Autoimmune disease (e.g., lupus erythematosis)
* Known allergic reactions or hypersensitivity to any of the components of the study preparations
* Allergy to adhesives on the patches used for occlusion in this study
* UV therapy in the four weeks before the study
* History of malignancy (except for treated or excised basal cell carcinoma)
* Surgery within the previous 3 months (except for minor cosmetic or dental procedures)
* History of drug or alcohol abuse (as defined by the Investigator)
* Symptoms of a clinically significant illness in the four weeks before the study that may influence the outcome of the study
* Positive for human immunodeficiency virus (HIV) antibody
* Systemic treatments in the two weeks preceding and during the study that may interact with any of the study drugs, such as: Glucocorticoids (po, im, iv), MAO inhibitors, Anti-depressants, Anti-seizure medications, Anti-psychotics, Antihistamines
* Subjects who require medications that inhibit the cytochrome P450 (CYP450) 2D6 pathway such as: Quinidine, Cimetidine, Type 1 antiarrhythmics, Phenothiazines, Selective serotonin reuptake inhibitors such as fluoxetine, paroxetine, and sertraline, reserpine, other anticholinergic drugs, and sympathomimetic drugs
* Participation in another clinical trial and/or treatment received with any investigational agent within one month before the initial dose of study medication
* Female subject who is pregnant or lactating
* Significant UV exposure in the four weeks before the study
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator or sponsor make the subject unsuitable for enrollment
* Subject is institutionalized because of legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Full skin thinning produced by treatment of CRx-191 in comparison with its components at corresponding dose levels, and vehicle with a marketed corticosteriod. Assess tolerability and safety of CRx-191. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gassmueller, M.D., Principal Investigator — Bioskin GmbH
Locations (1):
- bioskin GmbH, Hamburg, Germany